CLINICAL TRIAL: NCT01124747
Title: An Open-Label Study to Evaluate the Disposition of 14C-Labeled ASP1585 in Healthy Male Volunteers
Brief Title: A Study to Assess the Systemic Disposition of ASP1585 After Administration of 14C-labeled Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 1585-CL-0011
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Healthy; Pharmacokinetics of ASP1585
Keywords: ASP1585; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP1585 and 14C-Labeled ASP1585 (Experimental)
  Interventions: Drug: ASP1585; Drug: 14C-Labeled ASP1585

INTERVENTIONS:
Drug: ASP1585 — Oral
Drug: 14C-Labeled ASP1585 — Oral

SUMMARY:
The objective of this study is to assess the systemic disposition of ASP1585 after oral administration of 14C-labeled drug in healthy male subjects.

DETAILED DESCRIPTION:
Subjects will receive study drug for 18 days with a radioactive dose of study drug given on Day 15. Blood, urine and feces will be collected to confirm recovery of radioactivity.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 32 kg/m2, inclusive and minimum body weight 45 kg
* Agrees to sexual abstinence or to use a highly effective form of birth control which includes a barrier method throughout the study
* In good health

Exclusion Criteria:

* History of any clinically significant disease
* History of bowel obstruction, swallowing disorders, gastrointestinal disorders, gastrointestinal surgery, actively bleeding hemorrhoids, or gastric/duodenal ulcers
* Irregular bowel habits (<1 bowel movement per day)
* Clinically significant illness within 30 days
* Received any drug or medicine (prescription or over-the-counter), including topical medications, complementary and alternative medicines and vitamin and mineral supplements within 14 days prior to the first dose of study drug
* Received any investigational medication during the last 30 days or 5 half-lives, whichever is longer, prior to screening
* Consumes >10 units of alcohol per week or history of alcoholism or drug/chemical abuse within past 2 years
* Smokes cigarettes or other nicotine-containing products
* Anticipates an inability to abstain from alcohol use for 48 hours prior to first dose of study drug or from grapefruit, Seville oranges, star fruit or products containing these items from 72 hours prior to first dose of study drug until end of study
* Positive drug or alcohol screen at Screening or Day -1
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or gamma-glutamyl transferase (GGT) value of >2x upper limit of normal at Screening or Day -1
* Known positive for human immunodeficiency virus (HIV), Hepatitis A, Hepatitis B or Hepatitis C
* Unwilling or unable to swallow large numbers of capsules
* Significant blood loss, donated one unit of blood or more, or received a transfusion of any blood or blood product within 60 days or donated plasma within 7 days prior to Day -1
* Known cumulative radiation exposure >5 rems for the whole body, active blood forming organs, ocular lens, and gonads, and >15 rems for other organs
* Has had nuclear medicine procedures, computed tomography scans, or significant x-rays (other than dental) within the past 12 months, has received radiolabeled material within the last 6 months, or has had significant occupational radiation exposure
* Has participated in a radiolabled study within the last 6 months or participated in more than one radiolabeled study within the last 12 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Excretion of radioactivity in urine | Day 15 and up to Day 24
Excretion of radioactivity in feces | Day 15 and up to Day 24

SECONDARY OUTCOMES:
Radioactivity assessment through analysis of blood samples | Day 15 and up to Day 24

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- Madison, Wisconsin, United States